CLINICAL TRIAL: NCT06592053
Title: Affecting Factors for the Incidence of Chronic Pain After Mastectomy
Brief Title: Affecting Factors for Chronic Pain After Mastectomy
Acronym: CPMP
Status: Recruiting | Type: Observational
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Berkant Demiray, Principal Investigator, Ankara Etlik City Hospital
Other Study IDs: AEŞH-BADEK-2024-414
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Mastectomy; Pain, Chronic; Pain, Acute; Breast Surgery; Breast Cancer Surgery
MeSH Terms: conditions — Chronic Pain; Acute Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Breast Cancer Surgery Pain — Factors affecting the occurrence of chronic pain in patients undergoing elective mastectomy surgery will be investigated.
  Other Names: Breast Cancer Surgery Chronic Pain

SUMMARY:
Chronic post-mastectomy pain (CPMP) is a significant issue affecting many women after mastectomy. Factors like age, treatment type, and pre-surgery pain can increase the risk of developing this condition. By evaluating these factors, CPMP can be prevented more successfully and treatment strategies can be developed. This study aims to investigate the factors contributing to CPMP and contribute to the existing literature on this important topic.

DETAILED DESCRIPTION:
Chronic post-mastectomy pain (CPMP) is a common condition and is a significant clinical problem with a prevalence reported in the literature of up to 50%. Approximately 10% of patients experience severe pain, which has a significant impact on their quality of life. Since mastectomy is a frequently performed procedure, this syndrome affects a large number of women. Therefore, it is important to better understand the factors associated with the development of persistent pain.

Several theories have been proposed regarding the development of CPMP, including increased peripheral nociceptor sensitivity (primary hyperalgesia) at the site of injury, central neuronal sensitivity (central hyperalgesia) in spinal and supraspinal regions innervating the injured area, and inflammatory changes triggered by the central nervous system. Recommended methods to prevent CPMP include careful dissection, reduction of inflammatory responses, and the use of minimally invasive surgical techniques to prevent peripheral and central neuronal sensitization.

Epidemiological studies-both retrospective and prospective-have identified some of these risk factors, such as younger age, chemotherapy, radiotherapy, and the presence of preoperative pain or severe acute postoperative pain. Unfortunately, there are few studies on this topic, and the literature needs further support.

The hypothesis in this study is that if investigator can identify the factors that increase chronic pain after mastectomy, investigator can take measures against these factors and reduce the development of chronic pain. Therefore, this study aims to identify the factors contributing to chronic pain after mastectomy.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-80
* BMI 18-35 kg/m2
* ASA (American Society of Anesthesiologists) Scoring I-II-III
* Elective mastectomy surgery
* Elective mastectomy and axillary dissection surgery
* Patients who will undergo general anesthesia
* Patients who agree to participate in the study and sign a form

Exclusion Criteria:

* Patients under 18 and over 80 years of age
* Patients who do not want to participate in the study
* Patients with chronic pain or chronic opioid use
* Patients with alcohol, substance or drug addiction
* Patients with a history of previous mastectomy
* Patients with limited cooperation such as dementia, psychiatric disorders
* Pregnant and breastfeeding patients will be excluded from the study
* Patients who cannot communicate in their native language will be excluded from the study

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-80 years, with an ASA classification of I-II-III and a body mass index (BMI) between 18-35 kg/m², who will undergo mastectomy surgery or mastectomy with axillary dissection, will be included in our study.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Self-leeds assessment of neuropathic symptoms and sign findings in 3rd months. | Postoperative 3rd month
  Patients; self-Leeds assessment of neuropathic symptoms and sign (S-LANSS) findings will be evaluated in the 3rd postoperative month. Patients with an S-LANSS score of 12 and above will be diagnosed with chronic neuropathic pain. In this scoring, the patient can get at least 0 points. He can get a maximum of 24 points. If the patient's score is 12 or above, the possibility of neuropathic pain is considered high.

SECONDARY OUTCOMES:
Short Form 12 questionnaire in the 3rd month | Postoperative 3rd month
  Short Form 12 questionnaire will be evaluated in the 3rd month to evaluate the quality of life of the patients.
Short Form 12 questionnaire in the 6th month | Postoperative 6th month
  Short Form 12 questionnaire will be evaluated in the 6th month to evaluate the quality of life of the patients
Self-leeds assessment of neuropathic symptoms and sign findings at 6th months | Postoperative 6th month
  Patients; self-Leeds assessment of neuropathic symptoms and sign (S-LANSS) findings will be evaluated in the 3rd postoperative month. Patients with an S-LANSS score of 12 and above will be diagnosed with chronic neuropathic pain. In this scoring, the patient can get at least 0 points. He can get a maximum of 24 points. If the patient's score is 12 or above, the possibility of neuropathic pain is considered high.
Acute pain score | Up to 24 hours after the operation
  Pain will be assessed at rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain). Pain assessment will be made at 0, 1, 24th hours in the postoperative period.

CONTACTS AND LOCATIONS:
Overall Officials: Musa ZENGİN, Associate Professor, Study Director — Ankara Etlik City Hospital
Locations (1):
- Ankara Etlik City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No